CLINICAL TRIAL: NCT07338461
Title: High Resolution Imaging OCT Pilot Study
Brief Title: High Resolution Imaging OCT Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg Engineering GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: R-2025-1
Record Dates: First submitted 2025-11-25; First posted 2026-01-13 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-11

CONDITIONS: Normal Eyes; Age Related Macular Degeneration; Diabetic Retinopathy; Eyes With Retinal Diseases
MeSH Terms: conditions — Macular Degeneration; Diabetic Retinopathy | interventions — Optical Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Investigational device R1 (Experimental): Imaging with the investigational device R1
  Interventions: Device: Autofluorescence Imaging; Device: Infrared reflectance imaging; Device: OCT imaging; Device: OCTA imaging
- HighRes OCT (Experimental): Imaging with the investigational device HighRes OCT
  Interventions: Device: Autofluorescence Imaging; Device: Infrared reflectance imaging; Device: OCT imaging; Device: OCTA imaging
- SPECTRALIS (Other): Imaging with the approved device SPECTRALIS
  Interventions: Device: Autofluorescence Imaging; Device: Infrared reflectance imaging; Device: OCT imaging; Device: OCTA imaging

INTERVENTIONS:
Device: Autofluorescence Imaging — Autofluorescence imaging with blue and green light and, multicolor imaging
Device: Infrared reflectance imaging — Infrared reflectance imaging, 30° Field of View
Device: OCT imaging — OCT Imaging Volume and Line Scans
Device: OCTA imaging — OCT Angiography, volume and SCOUT scan

SUMMARY:
The goal of this pilot study is to compare image quality between the investigational devices (R1 and HighRes OCT) and the SPECTRALIS (cleared) in adult participants with normal and/or pathology eyes.

Participants will be imaged with different imaging modalities and scan protocols on all study devices.

ELIGIBILITY:
Inclusion Criteria:

* All Able and willing to undergo the test procedures, give consent, and to follow instructions.

Signed informed consent Age ≥ 18 years

* Healthy Subjects without uncontrolled systemic conditions, as determined by the investigator Subjects without ocular disease, as determined by the investigator Corrected visual acuity ≥ 20/40 No reported history of ocular surgical intervention (except for refractive or cataract surgery)
* Age-related macular degeneration Subjects with a diagnosis of AMD as determined by the investigator, either early-intermediate, atrophic, or neovascular
* Diabetic retinopathy Subjects with a diagnosis of diabetic retinopathy as determined by the investigator
* Disease with expected altered autofluorescence pattern Subjects with a disease that can be expected to be associated with altered autofluorescence patterns as determined by the investigator

Exclusion Criteria:

* Subjects unable to read or write
* Subjects with ocular media not sufficiently clear to obtain acceptable study-related imaging
* Subjects who cannot tolerate the imaging procedures
* History of photosensitive epilepsy
* Vulnerable subjects, i.e., individuals with lack of or loss of autonomy due to immaturity or through mental disability, persons in nursing homes, impoverished persons, subjects in emergency situations, homeless persons, nomads, refugees, and those incapable of giving informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
cSLO Image quality grading | 6 months after image acquisition
  Good: Good focus, even illumination, optimal exposure Average: The image is of sub-optimal quality, where there are issues with focus, illumination, or exposure, but the image still allows assessment of clinically relevant content Poor: Clinically relevant features are not visible, images are not clinically useful
Visability of key anatomical structures | 6 months after image acquisition
  Visibility of
  OCT image:
  1. Difference in reflectivity between the outer retino-choroidal complex and vitreous
  2. The vitreo-retinal interface
  3. Difference in reflectivity between retinal nerve fiber layer and vitreous
  4. Difference in reflectivity between plexiform layer and vitreous
  5. Multiple layers within the outer retino-choroidal complex
  6. The ganglion cell layer
  7. Difference in reflectivity between outer nuclear layer and vitreous
  8. External limiting membrane
  9. Choroidal/scleral interface
  OCTA image:
  1. Foveal avascular zone
  2. Large vessels: 1st order vasculature, if applicable
  3. Medium vessels: 2nd and 3rd order vasculature
  4. Small vessels: between 3rd order vasculature and end capillaries
  5. End capillaries

SECONDARY OUTCOMES:
Safety Monitoring | from enrollment to study completion (expected 1 year after initiation)
  Observation of possible adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Cozzi, MD, Principal Investigator — University of Milan, Department of Biomedical and Clinical Sciences, Luigi Sacco Hospital
Locations (1):
- Department of Biomedical and Clinical Sciences, Luigi Sacco Hospital, University of Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: No